CLINICAL TRIAL: NCT05550649
Title: Safety and Efficacy of Prophylactic Arterial Embolization in the Treatment of Angiography-negative Acute Upper Gastrointestinal Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Shilong Han, MD, Principal Investigator, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHSY-IEC-5.0/22K8/P01; 20204Y0167 (Other Grant/Funding Number: Shanghai Municipal Health Commission)
Record Dates: First submitted 2022-09-10; First posted 2022-09-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Acute Gastrointestinal Bleeding
MeSH Terms: interventions — Embolization, Therapeutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylic Embolization (Experimental): Prophylactic arterial embolization is performed for the artery in the diseased blood supply area. The embolization material: gelatin sponge particles are recommended, and micro-steel ring can be used as an auxiliary if necessary; after operation, symptomatic and supportive treatment such as acid suppression, hemostasis, blood transfusion, and fluid replacement are given according to the condition.
  Interventions: Procedure: embolization
- Sham Embolization (Sham Comparator): After the angiography was completed, no embolization was performed, the catheter was withdrawn, the vascular sheath was removed, and symptomatic and supportive treatments such as acid suppression, hemostasis, blood transfusion, and fluid replacement were given.
  Interventions: Procedure: embolization

INTERVENTIONS:
Procedure: embolization — Prophylactic arterial embolization is performed for the artery in the diseased blood supply area. The embolization material: gelatin sponge particles are recommended, and micro-steel ring can be used as an auxiliary if necessary; after operation, symptomatic and supportive treatment such as acid suppression, hemostasis, blood transfusion, and fluid replacement are given according to the condition.

SUMMARY:
Guided by clinical problems, this study focused on the problems encountered in clinical practice, with the interventional treatment of emergency gastrointestinal bleeding as the breakthrough point, and focused on the dilemma of treatment selection for patients with negative angiography in gastrointestinal bleeding. At present, there is no report on relevant clinical and basic research on the selection of treatment strategies for patients with negative ANVUGIB angiography. Whether prophylactic arterial embolization can benefit patients and whether it can reduce mortality is an urgent clinical problem to be solved.

DETAILED DESCRIPTION:
1. Research subjects Patients who were admitted to our hospital from January 2021 to December 2023 and underwent interventional therapy for acute non-variceal upper gastrointestinal bleeding and were negative on angiography were selected.

   Once the subjects signed the informed consent and participated in the screening, the subjects who met all the following inclusion criteria according to the experimental protocol and did not meet any of the exclusion criteria were eligible for screening.
2. Study endpoints 1) The primary endpoint: postoperative rebleeding rate. 2) Secondary endpoints: hemoglobin, hematocrit, blood transfusion volume, complication rate, mortality, surgical intervention rate.
3. In/Out Criteria 1) Inclusion criteria: (1) Age: 18~75 years old (including 18 years old and 75 years old); (2) Bleeding of gastric or duodenal ulcers that have failed endoscopic therapy; (3) Anastomotic bleeding after gastrointestinal anastomosis; (4) Anastomotic bleeding after cholangioenterostomy; (5) Bleeding after ERCP; (6) There were no indirect signs of contrast agent spillage and bleeding in angiography.

2) Exclusion criteria:

(1) Age: <18 years old or >75 years old; (2) Rupture and bleeding of gastric fundus esophageal varices; (3) Active bleeding can be seen on angiography; (4) Upper gastrointestinal bleeding caused by other causes other than the inclusion criteria; (5) Unexplained upper gastrointestinal bleeding; (6) Those who have undergone interventional therapy in the past; (7) Allergy to iodine-containing contrast agents; (8) Uncorrectable coagulation dysfunction and uncontrolled systemic infection; (9) There is functional failure of important organs (heart, liver, kidney, etc.); (10) History of gastrointestinal radiotherapy in the past 1 year; (11) Those who are not expected to complete the follow-up; (12) Expected survival shorter than 6 months. 3) Elimination criteria

1. After enrollment, it is found that the subjects do not meet the inclusion criteria or meet the exclusion criteria;
2. Other diseases or conditions occurred during the trial, which, as judged by the investigator, significantly affected the evaluation of clinical status and research endpoints;
3. Those whose treatment was interrupted due to various reasons or whose case records were incomplete, were determined by the investigators to be unevaluable.

4) Exit/Abort:

1. The subject himself or his legal representative requests to withdraw from the research;
2. Lost to follow-up;
3. DEATH. For all cases of rejection, withdrawal/discontinuation, the reason for rejection, withdrawal/discontinuation must be recorded on the case report form and subject medical records.

4. Interventional treatment process

1. Preoperative preparation: perfect electrocardiogram, gastroscope (optional), chest X-ray/chest CT (optional), enhanced abdominal CT (optional), blood routine, biochemistry, coagulation function, stool routine + occult blood, eight items before surgery etc.; signed informed consent for interventional therapy.
2. Angiography: (1) Prepare the skin at the puncture site, sterilize and lay down sheets; (2) Determine the puncture point: routinely choose the right femoral artery, or the left femoral artery or radial artery, (3) Lidocaine Anesthetize the puncture point, puncture and introduce the 4-5F arterial sheath; (4) Conventional angiography: celiac artery (5-7ml/s, total amount of contrast agent 25-35ml, 300 psi), superior mesenteric artery (5-7ml/s, Total volume of contrast agent 25-35ml, 300 psi). (5) Superselective angiography: superselective angiography of the blood supply artery in the lesion area is performed according to the cause of bleeding, the lesion site determined by endoscopic or enhanced CT, and the flow rate of contrast agent, the duration of angiography and the pressure are determined according to the diameter of the blood vessel.
3. Group processing:

(1) Control group: After angiography, no embolization was given, the catheter was withdrawn, the vascular sheath was removed, and symptomatic and supportive treatments such as acid suppression, hemostasis, blood transfusion, and fluid replacement were given.

(2) Observation group: Prophylactic arterial embolization was performed for the artery in the blood supply area of the lesion. Embolization material: gelatin sponge particles are recommended, and micro-steel ring can be used as an auxiliary if necessary; postoperatively, according to the condition, symptomatic acid suppression, hemostasis, blood transfusion, and fluid replacement were given. and supportive care.

Indications for blood transfusion: (1) systolic blood pressure < 90 mmHg, or a decrease of > 30 mmHg from baseline systolic blood pressure; (2) hemoglobin < 70 g/L, hematocrit < 25%; (3) increased heart rate (> 120 times/min).

4. Postoperative treatment: (1) Monitoring vital signs; (2) On the 1st, 7th, and 14th days after operation, and in January and March respectively, test blood routine, coagulation function, liver and kidney function, stool routine + occult blood, etc.; ( 3) Observe the bleeding situation; (4) Observe and record adverse reactions.

6. Angiographic findings

1. Positive signs of bleeding: contrast agent spillage, pseudoaneurysm, irregular arterial stenosis/truncation.
2. Negative signs of bleeding: the shape of blood vessels is obviously abnormal, and the above positive signs are not present on angiography.

6. Efficacy evaluation Technical success: Successful embolization of the target arterial vessel. Technical failure: The target artery was not successfully embolized. Clinical success: no more active bleeding within 1 month after surgery, or significant reduction in bleeding volume, no need for blood transfusion therapy Bleeding stopped: (1) bleeding from gastric tube or abdominal drainage tube stopped; (2) the patient's symptoms improved, heart rate and blood pressure were stable; (3) urine output > 0.5 ml/kg/h. Active bleeding: (1) bleeding from gastric tube or abdominal drainage tube; (2) increased frequency of hematemesis or melena, bright red vomit or dark red blood in stool, or active bowel sounds; (3) rapid infusion Blood transfusion, the performance of peripheral circulatory failure did not improve significantly, or although it temporarily improved and then deteriorated, the central venous pressure still fluctuated, stabilized and then decreased again; (4) red blood cell count, hemoglobin concentration and hematocrit continued to decline, reticulum The red blood cell count continued to increase; (5) the blood urea nitrogen continued or increased again when the fluid and urine volume were sufficient.

7. Safety evaluation:

1. Serious complications: require surgical treatment or prolong hospital stay for ≥2 weeks.
2. Mild complications: no surgical treatment or prolonged hospital stay is required for less than 2 weeks.

Recording of complications: from the time the subjects signed the informed consent, until the subjects completed or withdrew from the trial. All adverse events that occurred during the trial must be recorded on a case report form. The contents of the records should include: the occurrence time, severity, duration, measures taken and outcomes of adverse events.

Technical difficulties: For the judgment of negative angiography, it is generally accepted that when the bleeding rate is lower than 15ml/min, the bleeding point cannot be found by DSA angiography, but it is also related to the pressure of the high-pressure syringe, the diameter of the blood vessel and the experience of the operator.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~75 years old (including 18 years old and 75 years old);
2. Bleeding of gastric or duodenal ulcers that have failed endoscopic therapy;
3. Anastomotic bleeding after gastrointestinal anastomosis;
4. Anastomotic bleeding after cholangioenterostomy;
5. Bleeding after ERCP;
6. There were no indirect signs of contrast agent spillage and bleeding in angiography.

Exclusion Criteria:

1. Age: <18 years old or >75 years old;
2. Rupture and bleeding of gastric fundus esophageal varices;
3. Active bleeding can be seen on angiography;
4. Upper gastrointestinal bleeding caused by other causes other than the inclusion criteria;
5. Unexplained upper gastrointestinal bleeding;
6. Those who have undergone interventional therapy in the past;
7. Allergy to iodine-containing contrast agents;
8. Uncorrectable coagulation dysfunction and uncontrolled systemic infection;
9. There is functional failure of important organs (heart, liver, kidney, etc.);
10. History of gastrointestinal radiotherapy in the past 1 year;
11. Those who are not expected to complete the follow-up;
12. Expected survival shorter than 6 months.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
postoperative rebleeding rate | 1 month
  No more active bleeding within 1 month after surgery, or the bleeding volume is significantly reduced, and no blood transfusion is required

SECONDARY OUTCOMES:
Hemoglobin | 1 month
  Hemoglobin count
blood transfusion volume | 1 month
  how much blood the patients need
complication rate | 1 month
  if there are any complications
mortality | 1 month
  number of patients dead within one month
surgical intervention rate. | 1 month
  patients need surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No